CLINICAL TRIAL: NCT02975817
Title: Preventing Inadvertent Hypothermia in Children Undergoing Elective Neurosurgery in Malawi - a Prospective Randomized Clinical Trial
Brief Title: Preventing Inadvertent Hypothermia in Paediatric Neurosurgery in Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Kamuzu University of Health Sciences (Other)
Responsible Party: Principal Investigator, Anders Christian Feyling, Principal investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: hypomalawi
Record Dates: First submitted 2016-11-24; First posted 2016-11-29 (Estimated); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Hypothermia
Keywords: pediatric, intraoperative, neurosurgery, inadvertent
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hibler's (Experimental): Insert description from protocol
  Interventions: Other: Hibler's
- Warm Air (Active Comparator): Insert description from protocol
  Interventions: Other: Warm Air

INTERVENTIONS:
Other: Hibler's — Passive body heat retention using multiple-layer tight wrapping of patient
  Arms: Hibler's
Other: Warm Air — Active, convective warming of patient using warm air blanket
  Arms: Warm Air

SUMMARY:
The investigators wish to undertake a randomized controlled non-inferiority trial to evaluate the ability of a simple and low-cost method (Hibler´s method of wrapping the patient in multiple insulating layers) to prevent intraoperative heat-loss in children undergoing neurosurgery under anesthesia in Malawi. The control group will be heated actively with the use of warm-air blankets. The aim of this study is to evaluate whether Hibler´s method can provide a cheap and technically simple way of adequately preserving the patients´ core temperature in the operating theatre in a resource-poor setting.

DETAILED DESCRIPTION:
Hypothermia in the perioperative setting is receiving increasing attention in anaesthetic and surgical care. The paediatric age group is arguably at increased risk and thus deserves more intensive focus.

The investigators wish to undertake a randomized controlled non-inferiority study in which two different modalities for preventing inadvertent intraoperative hypothermia are compared. The trial will be carried out in a paediatric neurosurgical population in a South-East African regional tertiary care hospital.

The primary objective is to determine whether a low cost and simple method can be as effective and safe as a more expensive and technically demanding method. The goal is to recruit 40 patients in each of the two study arms. Patients younger than 12 years of age presenting for scheduled neurosurgery will be approached and given information about the study. If informed consent (and assent, where applicable) is obtained, participants will be randomized to one of the two different techniques; either passive heat preservation using what has become known as Hibler´s method (interventional group) or active warming with warm-air blankets (control group). Throughout the study period core temperature will be measured continuously, both for purposes of data accuracy and to maintain safety standards.

Primary study outcomes focus on the comparative ability of the methods in maintaining acceptable core temperatures. The trial will also examine a number of secondary end-points such as prevalence of shivering, conscious level, analgesia requirements, oxygenation and overall cost.

Upon completion of the study the investigators will seek to publish the findings in a relevant medical journal. Presenting the results in abstract form or as a poster in an appropriate medical congress may also be desirable.

ELIGIBILITY:
Inclusion criteria:

I. Age under 12 years. II. Ensured bed in HDU for postoperative management. III. Undergoing general anaesthesia with endotracheal intubation for planned cranial procedures; e.g. craniotomies, ventriculo-peritoneal shunt placements, endoscopic third ventriculostomies and similar procedures with a predominantly cranial access.

IV. Informed parental/guardian consent given

Exclusion criteria:

I. Pts. aged 12 years or older. II. Pts. with a temperature upon arrival at the anaesthetic suite lower than 36,0 °C III. Pts. with a temperature upon arrival at the anaesthetic suite greater than 37,5°C IV. Pts. judged to be unsuited for the standardized anaesthetic technique chosen (due to known allergy, known or suspected difficult airway requiring other anaesthetic interventions, cardiovascular conditions incompatible with the standard anaesthetic agents or due to any other condition where the chosen technique is deemed unsafe)

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2016-06; Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
incidence of hypothermia | from start of surgery till end of surgery
  incidence of core temperatures below 36,0 C

SECONDARY OUTCOMES:
incidence of postoperative shivering | postoperative period, from start of stay at HDU (High Dependency Unit) till 5 hours into this stay
  incidence of shivering at arrival at and at the end of the fifth hour of stay in HDU
Oxygen requirements | postoperative period, from start of stay at HDU (High Dependency Unit) till 5 hours into this stay
  requirement of supplemental oxygen (and mode of delivery) to maintain peripheral oxygen saturation at 95% or above
Degree of alertness | postoperative period, from start of stay at HDU (High Dependency Unit) till 5 hours into this stay
  Degree of alertness (as judged using a simple 5 step scale) at arrival at and at the end of the fifth hour of stay in HDU
Proportion of surgery time spent normothermic | from start of surgery till end of surgery
  proportion of surgery time spent at core temperature at or above 36,0 C

CONTACTS AND LOCATIONS:
Overall Officials: Anders C Feyling, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Queen Elizabeth Central Hospital, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Feyling AC, Kamalo PD, Hanche-Olsen T, Chikumbanje SS, Zsidek AS, Ponzi E, Raeder J. Preventing hypothermia in pediatric neurosurgery in Africa-A randomized controlled non-inferiority trial of insulation versus active warming. Acta Anaesthesiol Scand. 2024 Feb;68(2):167-177. doi: 10.1111/aas.14341. Epub 2023 Oct 26. PMID 37882145